CLINICAL TRIAL: NCT05858463
Title: Mitochondrial Adaptations and Oxidative Stress With High Intensity Interval Training During Pulmonary Rehabilitation
Brief Title: High Intensity Interval Training and Muscle Adaptations During PR
Acronym: MITOXITRAIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AOI 2022 COSTES; 2022-A02468-35 (Other: ANSM)
Record Dates: First submitted 2023-04-27; First posted 2023-05-15 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Mitochondrial Alteration; Oxygen Deficiency
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypoxia

STUDY DESIGN:
Intervention Model Description: comparison of 2 exercise training strategies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): High Intensity Interval training: 1 min at maximal workload followed by 1 min rest, repeated during a maximum of 40 min.
  Interventions: Other: Modality of exercise training
- Control group (Active Comparator): Low intensity continuous exercise training set at the level of the ventilatory threshold, lasting for a maximum of 40 min
  Interventions: Other: Modality of exercise training

INTERVENTIONS:
Other: Modality of exercise training — muscle adaptations following intermittent high intensity interval exercise training and continuous low intensity exercise training

SUMMARY:
Pulmonary rehabilitation (PR) is a validated treatment in patients with Chronic Obstructive Pulmonary Disease (COPD), improving exercise tolerance, quality of life and dyspnea. However, 20 to 30% of patients did not respond to PR and particularly those with chronic hypoxaemia. In most disabled patients, High Intensity Interval training (HIIT) is an alternative to perform exercise training with similar gain in exercise capacity than continuous exercise training. In patients with exercise-induced oxygen desaturation, the repetitions of hypoxia/resaturation phases during intermittent exercise could result in bursts of oxidative stress and induce positive or detrimental effect on mitochondrial function according to the importance in the oxidant stimulus.

Few data have ascertained the benefit of HIIT on mitochondrial oxidative capacity (Vmax) in healthy subjects compared to continuous exercise training but no data are available in COPD patients with exercise-induced desaturation, and the change in oxidative stress in such training regimen.

The investigators hypothesize that the repetitive bursts of oxidative stress and the improved antioxidant capacity in the course of the training sessions would stimulate mitochondrial adaptations to a larger extent after HIIT than continuous exercise training in severe COPD patients with hypoxemia. Moreover, they will assess the relationship between the change in oxidative stress in blood and in muscle. The clinical relevance of this study will be to ascertain the benefit and the safety of HITT in this subgroup of COPD patients in whom benefit of PR is often weak.

DETAILED DESCRIPTION:
The investigators will conduct an open-label randomized controlled trial in 2 parallel groups of COPD patients referred for a pulmonary rehabilitation programme (PR). After inclusion the patients will be randomized in HIIT (IG) or continuous groups (CG). Two visits will be planned before and 2 immediately after completion of PR, with similar tests.

1. A cycling endurance test performed until exhaustion CG: exercise at 75% of predetermined maximal workload (Wmax) IG: 1 min at Wmax followed with 1 min unloaded pedaling, up to a maximal duration of 30 minutes. During this test, oxygen consumption, minute ventilation, cardiac output (thoracic impedance), pulse oxygen saturation and muscle oxygen saturation (NIRS) will be recorded continuously.

   Markers of oxidative stress will be measured before and at the end of the cycling test (5 ml blood).
2. The mitochondrial oxidative capacity of the quadriceps will be measured on a separate day. A 20 mg biopsy of the vastus lateralis will be obtained under local anaesthesia using a biopsy needle. Maximal mitochondrial oxygen consumption (Vmax) will be measured on fresh permeabilized fibers (10 mg) using high resolution respirometry (Oroboros®), and 10 mg will be frozen for determination of oxidative markers. Vmax was also determined non invasively by the recovery of muscle oxygen saturation (NIRS) during repetitive brief arterial occlusions (according to the method described by Ryan and coll).

As part of PR, the participants will complete 20 sessions of exercise training (HIIT or continuous). The exercise intensity will be adapted weekly according to the participant's sensation. In the IG, the sessions will not exceed 40 min (20 min of active exercise).

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosed according to Global Obstructive Lung Diagnosis criteria; no exacerbation of COPD in the last month
* Referred for a pulmonary rehabilitation program
* Exercise-induced oxygen desaturation during a CardioPulmonary Exercise Test, defined as a decrease of oxygen saturation by pulse oximetry >4% from resting value.
* Written informed consent
* Negative pregnancy test whenever applicable.

Exclusion Criteria:

* Acute exacerbation of COPD during the last 4 weeks
* Physical or psychological inability to perform exercise tests
* Life-threatening cardiac events contra-indicating exercise training
* Anticoagulant treatment (muscle biopsy)
* Pregnant or breastfeeding womenFemmes
* Subject with curator, deprived of freedoms or in safeguard of justice
* Non covered by the french social security system

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Vmax variation | from the beginning to the end of the exercise training program (maximum duration 3 months)
  variation of maximal mitochondrial O2 consumption ( pmol O2.s-1.mg-1) ( with exercise training in both groups

SECONDARY OUTCOMES:
blood oxidative stress variation | from the beginning to the end of the exercise training program (maximum duration 3 months)
  variation with exercise training in both groups of blood oxidative stress, with a composite score obtained by the plasmatic levels of superoxide dismutase, gluthation peroxydase, xanthine oxidase, catalase and myeloperoxidase
mVO2 variation | from the beginning to the end of the exercise training program (maximum duration 3 months)
  variation of muscle oxidative capacity measured by NIRS(affinity constant, min-1) with exercise training in both groups
Cardiac output variations | from the beginning to the end of the exercise training program (maximum duration 3 months)
  variations with exercise training in both groups of cardiac output (L.min-1) measurements during endurance cycling exercise
Respiratory variations | from the beginning to the end of the exercise training program (maximum duration 3 months)
  variations with exercise training in both groups of minute ventilation (L.min-1) measurements during endurance cycling exercise
muscle oxygen variations | from the beginning to the end of the exercise training program (maximum duration 3 months)
  variations with exercise training in both groups of tissue index oxygenation (TIO,%) measured by Near Infrared Spectroscopy during endurance cycling exercise

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Costes, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France